CLINICAL TRIAL: NCT01615796
Title: A Two-Part Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Repeat IV Doses of GSK2140944 in Healthy Adult Subjects.
Brief Title: Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Repeat IV Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 115198
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infections, Respiratory Tract
Keywords: GSK2140944; antibiotics; first time in human; pharmacokinetics; intravenous; safety; absolute bioavailability; Bacterial Type II; tolerability; infection
MeSH Terms: conditions — Respiratory Tract Infections; Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (12):
- Cohort A1 (Experimental): GSK2140944 200mg single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort A2 (Experimental): GSK2140944 600mg single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort A3 (Experimental): GSK2140944 1200mg single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort A4 (Experimental): GSK2140944 1800mg single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort A5 (Experimental): GSK2140944 1800mg single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort A6 (Experimental): GSK2140944 dose to be determined, single dose
  Interventions: Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined
- Cohort B1 (Experimental): GSK2140944 400 mg repeat dose BID up to 7 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined
- Cohort B2 (Experimental): GSK2140944 750 mg repeat dose BID up to 7 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined
- Cohort B3 (Experimental): GSK2140944 1000 mg repeat dose BID up to 7 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined
- Cohort B4 (Experimental): GSK2140944 to be determined repeat dose BID up to 7 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined
- Cohort B5 (Experimental): GSK2140944 to be determined repeat dose TID up to 14 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined
- Cohort B6 (Experimental): GSK2140944 to be determined repeat dose TID up to 14 days
  Interventions: Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined

INTERVENTIONS:
Drug: Part A: GSK2140944 Drug single dose of 200mg, 600mg, 1200mg, 1800 mg, and dose to be determined — Subjects receive a single dose of GSK2140944
  Arms: Cohort A1; Cohort A2; Cohort A3; Cohort A4; Cohort A5; Cohort A6
Drug: Part B: GSK2140944 Repeat Drug dose of 400mg, 750mg, 1000 mg, and dose to be determined — Subjects will receive repeat doses of GSK2140944 BID/TID for up to 14 Days
  Arms: Cohort B1; Cohort B2; Cohort B3; Cohort B4; Cohort B5; Cohort B6

SUMMARY:
GSK2140944 belongs to the Bacterial Type II Topoisomerase Inhibitor (BTI) class of antibiotics. GSK2140944 has demonstrated in vitro and in vivo activity against Gram positive pathogens including methicillin resistant Staphylococcus aureus (MRSA) and Gram-negative pathogens associated with respiratory tract, skin and soft tissue infections including isolates resistant to existing classes of antimicrobials.

DETAILED DESCRIPTION:
GSK2140944 belongs to the Bacterial Type II Topoisomerase Inhibitor (BTI) class of antibiotics. GSK2140944 has demonstrated in vitro and in vivo activity against Gram positive pathogens including methicillin resistant Staphylococcus aureus (MRSA) and Gram-negative pathogens associated with respiratory tract, skin and soft issue infections including isolates resistant to existing classes of antimicrobials. This study will be the first administration of GSK2140944 as an intravenous (IV) formulation in humans and will be conducted in two (2) parts. Single IV doses will be explored in Part A and repeat IV doses will be explored in Part B. In addition, this study will evaluate the absolute bioavailability of an oral capsule formulation as compared to the IV formulation in Part A. Both study parts will investigate the safety, tolerability and pharmacokinetic profile of GSK2140944 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin less than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. To confirm post-menopausal status, a blood sample for simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the final follow-up visit.
* Body weight greater than and equal to 50 kg and BMI within the range 19 - 31 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or positive Human Immunodeficiency Virus (HIV) antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening.
* A screening urinalysis positive for protein or glucose (greater than "trace" findings of protein or glucose).
* A serum creatinine value between screening and Day -1 visit that is increased by more than 0.2 mg/dL (or 15.25 umol/L) changes.
* History of photosensitivity to quinolones.
* Unwillingness to commit to avoid excessive exposure to sunlight (or exposure whilst on a tanning bed) which would cause a sunburn reaction from first dose up to and including the follow-up visit.
* History of drug abuse within 6 months of the study.
* History of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units (or an average daily intake of greater than 3 units) for males or an average weekly intake of greater than 14 units (or an average daily intake greater than 2 units) for females. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take paracetamol or acetaminophen (less than and equal to 2 grams/day) up to 48 hours prior to the first dose of study medication. However, the Investigator and GSK study team can review medication on a case by case basis to determine if its use would compromise subject safety or interfere with the study procedures or data interpretation.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Donation of blood in excess of 500 mL within 12 weeks prior to dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of tendon rupture.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices containing such products from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate: Males - less than 40 and greater than 100 bpm; Females: less than 50 and greater than 100 bpm; PR Interval: Males and Females - less than 120 and greater than 220 msec; QRS duration: Males and Females - less than 70 and greater than 100 msec; QTcB or QTcF interval: Males and Females - greater than 450 msec; Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization); Subject has Bundle Branch Block; Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses greater than 3 seconds, non-sustained or sustained ventricular tachycardia (greater than and equal to 3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.
* Screening holter monitoring shows one or more of the following: Any symptomatic arrhythmia (except isolated extra systoles); Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, SVT (greater than 10 consecutive beats)); Sinus tachycardia (or supraventricular tachycardia) greater than 150 bpm; Non-sustained or sustained ventricular tachycardia (defined as greater than and equal to 3 consecutive ventricular ectopic beats); Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher in an awake subject], WPW syndrome, other pre-excitation syndromes); Symptomatic sinus pause or sinus pause >3 seconds - unless patient is straining, vomiting, or having some other type of hypervagal response; 300 or more supraventricular ectopic beats in 24 hours; 250 or more ventricular ectopic beats in 24 hours; Ischemia, diagnosed by a sequence of EKG changes that include flat or downsloping ST-segment depression greater than 0.1 mV, with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule).
* Neutrophil count <2000 cells per microliter (a single repeat is allowed for eligibility determination).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2014-02-21 (Actual); Study Completion 2014-02-21 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters of GSK2140944 including area under the curve following single dose administration. | Part A up to 4 days
  Measurements include area under the plasma concentration curve (AUC) from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity), AUC over the dosing interval AUC(0-tau). AUC (0-12) and AUC(0-24).
Composite of PK parameters for GSK2140944 following single dose administration | Part A up to 4 Days
  Measurements include maximum observed concentration (Cmax), systemic clearance of parent drug (CL). volume of distribution at steady state of parent drug after intravascular administration (Vdss), Mean residence time (MRT) and terminal phase half-life (t1/2)
Composite of PK parameters for GSK2140944 including area under the curve following repeat dose administration. | Part B Days 4, 7, 10 and 14
  Measurements include AUC from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity), AUC over the dosing interval AUC(0-tau). AUC (0-8), AUC (0-12) and AUC(0-24).
Composite of PK parameters for GSK2140944 following repeat dose administration. | Part B Days 4, 7, 10 and 14
  Measurements include Cmax, CL. Vdss, MRT and t1/2.
Composite of PK parameters for GSK2140944 following repeat dose administration including maximum concentration, area under the curve, accumulation ratio and clearance of parent drub. | Part B Days 4, 7, 10 and 14
  Measurements include AUC(0-tau). Cmax, pre-dose (trough) concentration at the end of the dosing interval (Cτ), accumulation ratio (Ro) and CL
GSK2140944 safety parameters - adverse events | Part A change from baseline for 15 Days. Part B change from baseline for up to 28 Days
GSK2140944 safety parameters - telemetry | Part A change from baseline for 15 Days. Part B change from baseline for up to 28 Days
GSK2140944 safety parameters - absolute values and changes over time of hematology, clinical chemistry and urinalysis | Part A change from baseline for 15 Days. Part B change from baseline for up to 28 Days
GSK2140944 safety parameters - vital signs (blood pressure, heart rate, temperature) | Part A change from baseline for 15 Days. Part B change from baseline for up to 28 Days
GSK2140944 safety parameters - Electrocardiogram (ECG) measurements | Part A change from baseline for 15 Days. Part B change from baseline for up to 28 Days

SECONDARY OUTCOMES:
A composite of pharmacokinetic parameters including dose proportionality following single and repeat doses of GSK2140944. | 44 Days in Part A, 7, 10 and 14 Days in Part B
  GSK2140944 AUC(0-∞) and Cmax for single doses and AUC(0-τ) and Cmax for repeat doses.
A composite of pharmacokinetic urinary parameters to estimate the urinary excretion of unchanged GSK2140944 following a therapeutically relevant dose and higher single dose in healthy volunteers. | 4 Days in Part A
  The amount of unchanged GSK2140944 in urine (Ae), fraction of the dose excreted in urine (fe) and renal clearance (CLr).
A composite of pharmacokinetic parameters to estimate the absolute bioavailability of the oral capsule formulation of GSK2140944 as compared to the IV formulation following single equivalent doses in healthy volunteers. | 4 Days in Part A
  Compare oral mean residence time (MRTpo), oral mean absorption time (MATpo) and absolute bioavailability of capsule formulation to IV formulation.
A composite of pharmacokinetic parameters to examine the extent of accumulation and time invariance following repeat doses of GSK2140944. | 4, 7, 10 and 14 days in Part B
  Measurements include Ro using AUC(0-τ) for repeat dose and AUC(0-12) for single dose, time invariance using repeat dose AUC(0-τ) and single dose AUC(0-∞)
A composite of pharmacokinetic parameters to examine achievement of steady-state following repeat doses of GSK2140944. | 7, 10 and 14 days in Part B
  Trough concentrations at the end of the dosing interval (Ctau) collected at pre-morning dose on Days 7 and 8 (together with pre-morning dose Ctau on Days 9 from the full PK profiles on Day 9) or Ctau collected at pre-morning dose on Days 10 and 11 (together with pre-morning dose Ctau on Day 12 from the full PK profiles on Day 12) or Ctau collected at pre-morning dose on Days 14 and 15 (together with pre-morning dose Ctau on Day 16 from the full PK profiles on Day 16) to assess achievement of steady-state.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115198 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115198?search=study&search_terms=115198#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register